CLINICAL TRIAL: NCT00340847
Title: Construction and Use of Lung Tumor Microarray for the Analysis of Gene Expression in Lung Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901233; 01-C-N233
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-19

CONDITIONS: Lung Cancer
Keywords: Molecular Profiling; In Situ Hybridization; SAGE; Tumor Markers; IHC; Lung Cancer; Genetics
MeSH Terms: conditions — Lung Neoplasms

SUMMARY:
The proposed research intends to construct a set of tissue microarrays containing different types of normal and lung cancer tissues for the study of genes associated with lung cancer. Thus far we have generated a lung cancer tissue arrayusing paraffin embedded archival tissues from 300 lung turmors tissues and 100 adjacent normal tissues. Four- micrometer thickness sections have been cut from the tissue array and were used to survey gene expression status in arrayed tumors using immunohistochemistry methody. We are currently performing IHC studies ot 1) determine protein expression and its correlation with gene expression patterms ovserved using cDNA arrays. 2) Analyze protein expression in the chromosome remodeling pathyway in non-small cell lung cancer. And 3) determine the association of gene expression with lung tumor stage and clinical outcome. The current protocol is needed to complete the above studies and for the production of neuroendocrine tumors.

DETAILED DESCRIPTION:
The proposed research intends to construct a set of tissue microarrays containing different types of lung cancer tissues for the study of genes associated with lung cancer. In this study, lung tissue arrays will be generated using paraffin embedded archival tissues containing adjacent normal tissues and tumors from approximately 300 non-small cell lung cancers and 100 neuroendocrine tumors of the lung. Corded tissues of 0.6 um in diameter will be taken from each tumor and arrayed onto recipient paraffin blocks to generate a lung tumor specific microarray. Four-micrometer thickness sections will be cut from the tissue array and used to survey gene expression status in arrayed tumors using fluorescence in situ hybridization (FISH, in situ hybridization, and/or immunohistochemistry methods. Additionally, approximately 20 sections will be cut from each primary tumor block to isolate genomic DNA for the analysis of genetic changes in the arrayed tumor samples. The goals of this proposal are 1) to generate a single tissue block containing multiple tumors, 2) allow rapid and efficient analysis of gene expressions in a large number of samples using a single tissue section, and 3) to correlate the molecular changes in the tumors with the clinical and pathological features of the disease. Due to the experimental nature of the research and the fact that all tumors obtained are archival tissues at AFIP, the investigators will not report the result of gene expression back to the subject.

To date, all samples needed for the protocol have been reached and there will be no more patient accrual but survival status of the patients as well as molecular analysis using the constructed lung tissue microarrays will continue for the foreseeable future.

ELIGIBILITY:
* INCLUSION CRITERIA

The human tissue microarrays will include existing archival tissues of normal lung, non small-cell lung cancer, and combined histological types of lung cancer samples. All tissue samples are already in existence at the Armed Forces Institute of Pathology.

The primary selection criteria will be the type of cancer, the quality of the tumor block, and the availability of the sample without regard to age, race, ethnic origin, and gender of the patient.

Only tissue blocks of suitable fixation quality and proper diagnosis will be used to generate the lung tissue microarrays.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2001-08-09; Study Completion 2010-05-19

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States